CLINICAL TRIAL: NCT06464757
Title: Laryngomalacia, Examinations and Quality of Life in Children Before and After Treatment With Follow-up After 1 Year
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Harriet Akre, Professor, Oslo University Hospital
Other Study IDs: 646948
Record Dates: First submitted 2024-05-21; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Laryngomalacia; Sleep Apnea, Obstructive; Sleep Apnea; Ear, Nose and Throat Disorder; Pediatric Disorder; Surgery; Quality of Life
MeSH Terms: conditions — Laryngomalacia; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with laryngomalacia
- Healthy children

SUMMARY:
Laryngomalacia is the most frequent cause of stridor in children under 1 year. The airway obstruction generates turbulent airway flow and creates the characteristic high-frequency stridor sound. In addition, the airway obstruction can cause apnea, a following drop in oxygen saturation and sleep disturbances. The symptoms of laryngomalacia are often worsened by activity, feeding, crying and lying flat on the back. The diagnosis is made with flexible laryngoscopy when the child is awake. The children are most often treated with expectation, information and guidance, observation with help with feeding and reflux treatment. Up to 20% of patients have a severe degree of laryngomalacia with apneas, which is an indication for surgical treatment. The investigators want to examine whether sleep examinations can help us deciding which child benefit from surgery, and follow-up the child again after 4-6 weeks and 1 year. The sleep examinations are carried out with polygraphy and/or polysomnography with simultaneous audio records and video monitoring and with Somnofy from VitalThings. The investigators want to use artificial intelligence and machine learning when analyzing the sleep examinations. The investigators also want to have a control group examining the sleep and breathing during night at home. In both groups the investigators want to examine the quality of life with the questionnaire ITQoL-SF47.

DETAILED DESCRIPTION:
Breathing difficulties in young children are a common cause of contact in the health care system, and are often related to harmless infection-triggered conditions in the upper and lower respiratory tract. In the vast majority of the cases, the condition is self-limiting and the child can be treated in primary care. In more serious or long-term cases, the child is referred to the specialist health care, most often to pediatricians, where the focus is naturally directed to pulmonary medical causes such as asthma, allergies and infections, as these make up the majority of breathing difficulties in children. Less common and less well-known are breathing difficulties in young children caused by airway obstructions in the upper airways, which might cause a characteristic respiratory distress called stridor. Stridor occurs as a result of turbulent airflow through a relatively narrower part of the upper airways, such as the larynx and trachea, and produces a high-frequency whistling sound during inspiration. Causes of stridor can be congenital or acquired, and stridor can often be confused with asthma. It is appropriate to refer to an ENT doctor for a thorough anatomical examination of the upper respiratory tract in these affected children to identify the cause of stridor and to be able to provide the correct treatment.

Laryngomalacia is the most frequent cause of stridor in children under 1 year of age, and is a congenital condition where the tissue at the top of the larynx collapses over the airway opening to the larynx and therefore creates an upper airway obstruction during inspiration. In severe cases, laryngomalacia can be curatively treated with surgery.

For long time the ENT departments and pediatric departments at regional hospitals in Norway have been responsible for the treatment of children under 1 year of age with laryngomalacia. However, experience in children under 1 year with laryngomalacia is limited, and there is a lack of systematic mapping and follow-up of these children. In Health South-East in Norway, with approximately 3.1 million inhabitants, children with a severe degree of stridor will be referred to the ENT department and/or the pediatric department at Oslo University Hospital. In addition, Oslo University Hospital also receives children with stridor from other health regions in Norway. Therefore, the patient base is well suited for a systematic mapping and follow-up. In this research project, the investigators want to carry out a mapping and follow-up of children with laryngomalacia, investigate how affected these children are by their breathing difficulties and the impact it has on sleep and quality of life on the child and the family. The investigators also want to investigate whether the treatment improves these variables.

In addition, the investigators want to recruit a control group of healthy children under 1 year of age to examine sleep and mapping the quality of life of the child and family. These children will be recruited from health centers, and the investigators want to follow them for up to 1 year.

In both groups the investigators want to use artificial intelligence and machine learning when analyzing the sleep examinations.

ELIGIBILITY:
Inclusion Criteria:

* laryngomalacia
* stridor
* breathing difficulties

Exclusion Criteria:

- none

Ages: 1 Week to 52 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with laryngomalacia, stridor and/or breathing difficulties.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea-index | 10 years
  Apnea-hypopnea-index
Quality of life in toddlers | 10 years
  Quality of life by using the Infant and Toddler Quality of Life Questionnaire (ITQOL-SF47)

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - Lovisenberg Diaconal Hospital, Oslo